CLINICAL TRIAL: NCT01376349
Title: Vaginal DHEA for Vaginal Symptoms: A Phase III Randomized, Double Blind, Placebo- Controlled Trial
Brief Title: Prasterone (Dehydroepiandrosterone) in Treating Postmenopausal Cancer Survivors With Vaginal Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N10C1; NCCTG-N10C1; CDR0000702003 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02677 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Gynecologic Cancer
Keywords: depression; anxiety disorder; cognitive/functional effects; sexual dysfunction; cancer survivor; breast cancer; cervical cancer; fallopian tube cancer; uterine sarcoma; vaginal cancer; vulvar cancer; ovarian epithelial cancer; ovarian germ cell tumor; ovarian sarcoma; ovarian stromal cancer; primary peritoneal cavity cancer; endometrial cancer
MeSH Terms: conditions — Breast Neoplasms; Depression; Anxiety Disorders; Sexual Dysfunction, Physiological; Uterine Cervical Neoplasms; Fallopian Tube Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Carcinoma, Ovarian Epithelial; Endometrial Neoplasms | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I low dose DHEA (Experimental): Participants apply a low dose (3.25 mg) of vaginal prasterone (dehydroepiandrosterone [DHEA]) gel once daily (QD), at bed time, for 12 weeks. Treatment continues until unacceptable adverse events or patient refusal to continue participation on the study.
  Interventions: Drug: prasterone
- Arm II high dose DHEA (Experimental): Participants apply a high dose (6.5 mg) of vaginal DHEA gel QD, at bed time, for 12 weeks. Treatment continues until unacceptable adverse events or patient refusal to continue participation on the study.
  Interventions: Drug: prasterone
- Arm III placebo (Placebo Comparator): Participants apply a vaginal placebo gel QD, at bed time, for 12 weeks. There is an Optional Continuation Phase (for placebo arm only): Participants apply a high dose of vaginal DHEA gel QD, at bed time, for 12 weeks. Treatment continues until unacceptable adverse events or patient refusal to continue participation on the study.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: prasterone — Applied vaginally
  Arms: Arm I low dose DHEA; Arm II high dose DHEA
Other: placebo — Applied vaginally
  Arms: Arm III placebo

SUMMARY:
RATIONALE: Dehydroepiandrosterone (DHEA) may help relieve vaginal symptoms in female cancer survivors.

PURPOSE: This randomized phase III trial studies DHEA to see how well it works compared to placebo in treating postmenopausal cancer survivors with vaginal symptoms.

DETAILED DESCRIPTION:
Primary Goal:

* To determine the effectiveness of two doses of daily vaginal prasterone (dehydroepiandrosterone [DHEA]) versus placebo for alleviation of the most bothersome vaginal symptom (vaginal dryness or dyspareunia) over 12 weeks.

Exploratory Goals:

* To evaluate any toxicities arising from DHEA in this patient population. (Exploratory)
* To evaluate the impact of vaginal DHEA on negative sexual thoughts, sexual function and urologic symptoms. (Exploratory)
* To explore the role of psychologic (mood, stress), physical (demographics and treatment variables) and situational factors (partner variables and fatigue) as predictors of vaginal dryness and performance outcomes at baseline and at various endpoints throughout the study. (Exploratory)
* To explore the characteristics of vaginal atrophy and the relationship between vaginal atrophy and quality-of-life questionnaire responses and exposure to hormonal therapy (tamoxifen, exemestane, anastrozole, or letrozole). (Exploratory)
* To examine the effects of the use of open-label vaginal DHEA gel over 8 weeks in women completing the placebo gel arm of the randomized trial. (Exploratory)

Correlative Research Goals:

* To evaluate the impact of vaginal DHEA on maturation index and pH (select institutions).
* To evaluate the impact of vaginal DHEA on sex steroid concentrations (estradiol, free testosterone, estrone, and DHEA-S) and markers of bone turnover (osteocalcin and bone alkaline phosphatase). (Correlative)
* As part of ongoing research for NCCTG Cancer Control studies, we are banking blood products for future studies. (Correlative)

OUTLINE: This is a multicenter study. Patients are stratified according to current tamoxifen therapy (yes vs no), concurrent aromatase inhibitor use (anastrozole/letrozole vs exemestane vs none), hysterectomy (yes vs no), and cigarette smoking (current vs past vs never). Patients are randomized to 1 of 3 treatment arms, patients receive low dose vaginal DHEA, high dose vaginal DHEA or vaginal placebo gel.

Participants may complete the Profile of Mood States (POMS), the Perceived Stress Scale (PSS), the Fatigue: Vitality subscale of the SF-36, the Vaginal Symptom Quality Questionnaire, the DHEA Side Effect Questionnaire, the Female Sexual Function Index (FSFI), the Sexually Related Intrusive Thoughts - ITS, Impact of Treatment Scale, the Urogenital Atrophy Questionnaire, and the Subject Global Impression of Change at baseline and periodically during study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Postmenopausal women with a history of breast or gynecologic cancer (currently no evidence of disease). Note: Postmenopausal status will be determined by the following criteria:

   1. 12 months without a period or bilateral oophorectomy or complete chemical ovarian suppression for the past 12 months with continued suppression planned throughout the course of the study
   2. menopausal status will be determined by an FSH and an estradiol value in the postmenopausal range (generally FSH > 40IU/L and estradiol < 10 pg/ml, depending on laboratory) if:

      * 9 months without a period or
      * post hysterectomy with at least one ovary remaining and less than 55 years old. Note: if age 55 or older with these criteria, then menopausal status does not need to be determined by labs
3. Significant vaginal complaints. Note: Defined as persistent vaginal dryness and/or pain with intercourse (dyspareunia) of sufficient severity to make a patient desire therapeutic intervention.
4. Eligibility questionnaire response must be moderate or worse levels of severity on one of the two symptoms, either dryness or dyspareunia. The protocol contains more information.
5. Vaginal symptoms must have been present ≥ 2 months prior to randomization.
6. Life expectancy > 12 months.
7. Ability to complete questionnaires by themselves or with assistance.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
9. The patient must provide informed written consent.
10. Willing to return to the enrolling institution for follow-up.
11. Willing to provide blood samples for correlative research purposes.

Exclusion Criteria:

1. Initiation or discontinuation of tamoxifen or aromatase inhibitors ≤ 2 months prior to randomization or plans to initiate or discontinue any of these medications during the 12-week study.
2. Current diagnosis of an active vaginal infection, if symptoms of vaginal infection, this must be ruled out (ie, foul discharge, fever).
3. Concurrent chemotherapy (long term adjuvant herceptin, lapatanib, and/or bevacizumab is allowed.
4. Planned use of any vaginal preparations during the study period (including any over the counter or herbal preparations). Note: Water-based lubricants (such as KY jelly) are allowed during sexual intercourse.
5. Use of any daily non-hormonal vaginal preparations ≤ 1 week prior to study entry.

   Exception: Daily water-based lubricants for sexual intercourse. Note: Patients who stop agent may be enrolled after one week.
6. Current (≤ 4 weeks prior to randomization), or planned during the study period, use of any estrogen product or any kind of hormonal vaginal product including bioidentical hormones, estriol or any androgen product.
7. Use of pharmacologic soy or phytoestrogen preparations (Dietary intake of soy - ie milk is acceptable).
8. On a placebo controlled trial for endocrine therapy.
9. Prior or concurrent pelvic radiation therapy.
10. Prior radical pelvic surgery, specifically vaginectomy or pelvic exenteration (TAH/BSO) is allowed).
11. Diagnosis of any of the following conditions within the past five years:

    1. Essential vulvodynia
    2. Vulvar vestibulitis
    3. Bartholin cyst/abscess
    4. History of Bartholin gland surgery
    5. Lichen sclerosis
    6. Lichen planus of the vulvovaginal region
    7. Desquamative vaginitis
12. History or current diagnosis of any of the following conditions:

    1. Vulvar or vaginal dysplasia
    2. Vaginal prolapse
13. Women of childbearing potential, premenopausal women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2011-07; Primary Completion 2013-08 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Barton, RN, PhD, AOCN, FAAN, Principal Investigator — University of Michigan
Locations (280):
- United States (280):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Herbert D. Kerman Regional Oncology Center - Daytona Beach, Daytona Beach, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Idaho Urologic Institute, PA, Meridian, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Francis Hospital Cancer Care Services, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Mercy Clinic Cancer and Hematology - Rolla, Rolla, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center - South, Las Cruces, New Mexico
  - Rutherford Hospital, Rutherfordton, North Carolina
  - MeritCare Broadway, Fargo, North Dakota
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Carolina Blood and Cancer Care Associates, PA, Lancaster, South Carolina
  - Carolina Blood and Cancer Care, Rock Hill, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 464 patients were accrued to this trial. Nineteen patients withdrew consent prior to randomization and were not included in the analysis of this study. Two additional patients were unable to classify the primary symptom and were not randomized to the trial and were not included in the analysis.
Period: Raondomized Treatment
Arm/Group | Arm I Low Dose DHEA | Arm II High Dose DHEA | Arm III Placebo
Started | 147 | 149 | 147
Completed | 123 | 114 | 118
Not Completed | 24 | 35 | 29
Not completed — Withdrawal by Subject | 10 | 16 | 13
Not completed — Adverse Event | 13 | 17 | 14
Not completed — Unkown | 1 | 2 | 1
Not completed — Alternative Treatment | 0 | 0 | 1
Period: Optional Continuation Phase
Arm/Group | Arm I Low Dose DHEA | Arm II High Dose DHEA | Arm III Placebo
Started | 0 | 0 | 94 (Patients completing Arm III Placebo were offered the option of continuing High Dose DHEA)
Completed | 0 | 0 | 94
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients that were randomized to treatment were included in baseline characteristics.
Groups:
- Arm III Placebo: Participants apply a vaginal placebo gel QD, at bed time, for 12 weeks. >
  > There is an Optional Continuation Phase (for placebo arm only): Participants apply a high dose of vaginal DHEA gel QD, at bed time, for 12 weeks. Treatment continues until unacceptable adverse events or patient refusal to continue participation on the study.
- Total: Total of all reporting groups
Arm/Group | Arm I Low Dose DHEA | Arm II High Dose DHEA | Arm III Placebo | Total
Number analyzed (Participants) | 147 | 149 | 147 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (6.7) | 57.3 (8.2) | 58 (7.3) | 57.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 149 | 147 | 443
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 147 | 149 | 147 | 443

OUTCOME MEASURES:

1. Primary Outcome: Alleviation of the Most Bothersome Vaginal Symptom (Vaginal Dryness or Dyspareunia) Over 12 Weeks
Description: The primary outcome is severity of the most bothersome vaginal symptom: dryness or dyspareunia. The Vaginal Symptom Measure (VSM) was used to evaluate the severity of vaginal dryness and dyspareunia. The VSM uses a 5- point ordinal response scale; 1="none", 2="mild", 3="moderate", 4="severe" and 5="very severe" to measure the severity associated with vaginal dryness and/or dyspareunia. For each patient, the change in severity was calculated by subtracting the baseline from the week 12 reported score. Therefore, the full range of scores ranges from -4 (greatest decrease in severity) to 4 (greatest increase in severity). A negative score indicates a decrease in severity from baseline, zero indicates no reported affect and positive scores indicate a more severe report at week 12. The primary assessment method will be a comparison of the averages of the changes over time in the severity items for the most bothersome symptom from baseline to 12 weeks (as indicated at baseline).
Time Frame: At baseline and 12 weeks
Population: All patients that started treatment and completed their week 12 evaluation are included in this analysis.
Measure: Median (Full Range); unit: change in units on a scale
Arm/Group | Arm I Low Dose DHEA | Arm II High Dose DHEA | Arm III Placebo
Number analyzed (Participants) | 123 | 114 | 118
change in units on a scale | -2 [-4 to 1] | -2 [-4 to 1] | -1 [-4 to 1]
Statistical Analysis 1: Comparison: Arm II High Dose DHEA vs Arm III Placebo; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I Low Dose DHEA vs Arm III Placebo; Test type: Superiority or Other; p = 0.48, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: All patients that started treatment and were assessed for adverse events were included in this section. This includes all 147 patients from Arm I, 148 patients from Arm II (one patient was not assessed for Adverse Events), and 147 patients from Arm III. In addition, patients from Arm III: Placebo were given the opportunity to receive treatment according to the Arm II: High Dose schedule upon completion of 12 weeks. 94 of the 147 patients randomized to Arm III opted to continue treatment.
Groups:
- Arm I: Low Dose DHEA: Participants apply a low dose (3.25 mg) of vaginal prasterone (dehydroepiandrosterone [DHEA]) gel once daily (QD), at bed time, for 12 weeks. Treatment continues until unacceptable adverse events or patient refusal to continue participation on the study.
- Arm II: High Dose DHEA: Participants apply a high dose (6.5 mg) of vaginal DHEA gel QD, at bed time, for 12 weeks. Treatment continues until unacceptable adverse events or patient refusal to continue participation on the study.
- Arm III: Placebo: Participants apply a vaginal placebo gel QD, at bed time, for 12 weeks.
  There is an Optional Continuation Phase (for placebo arm only): Participants apply a high dose of vaginal DHEA gel QD, at bed time, for 12 weeks. Treatment continues until unacceptable adverse events or patient refusal to continue participation on the study.
- Optional Continuation Phase: Patients randomized to Arm III Placebo who have completed protocol treatment for 12 weeks were offered the option of continuing treatment according to Arm II High Dose DHEA until unacceptable adverse events or patient refusal to continue participation on the study.
  94 of the 147 patients randomized to the Placebo arm opted to continue treatment with High Dose DHEA.
Arm/Group | Arm I: Low Dose DHEA | Arm II: High Dose DHEA | Arm III: Placebo | Optional Continuation Phase
Serious Adverse Events (participants affected / at risk) | 3/147 | 7/148 | 4/147 | 0/94
Other Adverse Events (participants affected / at risk) | 91/147 | 105/148 | 93/147 | 28/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Low Dose DHEA (N=147) | Arm II: High Dose DHEA (N=148) | Arm III: Placebo (N=147) | Optional Continuation Phase (N=94)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Low Dose DHEA (N=147) | Arm II: High Dose DHEA (N=148) | Arm III: Placebo (N=147) | Optional Continuation Phase (N=94)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestine ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (2) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 5 (6) | 3 (3) | 2 (5) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Breast infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urethral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (9) | 3 (3) | 5 (5) | 0 (0)
Vaginal infection (Infections and infestations) | 3 (6) | 5 (6) | 2 (3) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 54 (130) | 55 (112) | 51 (145) | 12 (18)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorgasmia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 29 (78) | 39 (96) | 33 (94) | 7 (14)
Dyspareunia (Reproductive system and breast disorders) | 2 (7) | 1 (1) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 6 (13) | 7 (9) | 5 (6) | 2 (3)
Vaginal dryness (Reproductive system and breast disorders) | 9 (33) | 4 (4) | 1 (1) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 1 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 8 (18) | 16 (32) | 15 (29) | 2 (2)
Hirsutism (Skin and subcutaneous tissue disorders) | 15 (50) | 26 (86) | 20 (50) | 6 (11)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 2 (2) | 10 (26) | 7 (13) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 12 (20) | 33 (56) | 27 (58) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (16) | 11 (14) | 12 (24) | 2 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less